CLINICAL TRIAL: NCT01222559
Title: Prospective, Randomised, Open Label, Multicentre Phase-III Clinical Trial to Compare the Efficacy and Safety of the Treatment With the Autologous Chondrocyte Transplantation Product co.Don Chondrosphere (ACT3D-CS) With Microfracture in Subjects With Cartilage Defects of the Knee With a Defect Size Between 1 an 4 cm2
Brief Title: Efficacy and Safety Study of co.Don Chondrosphere to Treat Cartilage Defects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: co.don AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: cod16HS13; 2009-016466-82 (EudraCT Number)
Record Dates: First submitted 2010-10-15; First posted 2010-10-18 (Estimated); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Articular Cartilage Lesion of the Femoral Condyle
Keywords: Cartilage defects; Knee joint; Femoral Condyle
MeSH Terms: interventions — Arthroplasty, Subchondral

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- co.don chondrosphere® (Experimental): co.don chondrosphere® are spheroids in suspension, developed from autologous chondrocytes. The dose depends on the size of the defect, recommended dose is 10-70 spheroids/cm2 defect.
  Interventions: Drug: co.don chondrosphere®
- Micofracture (Active Comparator): A procedure in which the subchondral bone is perforated to allow a bloodcloth to form scar tissue.
  Interventions: Drug: co.don chondrosphere®; Procedure: Microfracture

INTERVENTIONS:
Drug: co.don chondrosphere® — co.don chondrosphere® are spheroids in suspension, developed from autologous chondrocytes. The dose depends on the size of the defect, recommended dose is 10-70 spheroids/cm2 defect.
  Other Names: ACT3D-CS
Procedure: Microfracture — A procedure in which the subchondral bone is perforated to allow a bloodcloth to form new tissue.
  Other Names: Subchondral drilling
  Arms: Micofracture

SUMMARY:
This is a prospective, phase III, multicenter, open label, randomised clinical trial of co.don chondrosphere®, a three-dimensional autologous chondrocyte transplantation product (ACT3D-CS)compared to the procedure of microfracture (MF)in the treatment of cartilage defects of knee joints.

After screening visit patients were booked for arthroscopy and at that time they were randomised to either ACT3D-CS with co.don chondrosphere® (Group A) or to MF(Group B), a marrow-stimulating method based on the penetration of the subchondral bone plate at the bottom of the cartilage defect. At the time of arthroscopy Patients of group B had their procedure of MF (treatment surgery) and patients of group A had their cells harvested from healthy cartilage. The cells are cultivated for 8-10 weeks in vitro to develope 3-dimensional spheroids , that are transplanted in an open knee procedure (treatment surgery)into the defect. Patients subsequently followed the same rehabilitation program and had post-surgery visits. After the 12-month-visit a interim analyses will be performed and the 24-month-visit is defined as final assessment. Then patients have follow-up assessments up to 60 months post-treatment-surgery.

DETAILED DESCRIPTION:
see above

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients, age: between 18 and 50 years
2. Defect: isolated ICRS grade III or IV single defect chondral lesions on femoral condyles
3. Defect size: 1 to < 4 cm2 after debridement to healthy cartilage up to 6 mm in depth.Assessment with MRI at screening and per estimation during arthroscopy prior to randomization
4. Nearly intact chondral structure surrounding the defect as well as an intact corresponding joint area
5. Informed consent signed and dated by patient
6. Patient understands the strict rehabilitation protocol and follow-up programme and is willing to follow it
7. In case of pain, patient agrees to use only paracetamol mono- (max 4 g/day) or combination preparation and oral and/or topic NSAIDs during the trial and to discontinue the use of oral and/or topic NSAIDs and/or paracetamol combination preparation 1 week before each visit whereas the use of paracetamol monopreparation (max 4 g/day) is allowed. However, in the morning of the visit day, no pain medication is allowed. Other pain medications are allowed during surgical procedure and may be taken for a period not exceeding 4 weeks after surgery.

Exclusion Criteria:

1. Defects on both knees at the same time
2. Radiological signs of osteoarthritis
3. Osteochondritis dissecans (OCD)
4. Any signs of knee instability
5. Valgus or varus malalignment (more than 5° over the mechanical axis)
6. Clinically relevant second cartilage lesion on the same knee
7. More than 50 % resection of a meniscus in the affected knee or incomplete meniscal rim
8. Rheumatoid arthritis, parainfectious or infectious arthritis, and condition after these diseases
9. Pregnancy and planned pregnancy (no MRI possible)
10. Obesity (Body Mass Index >30)
11. Uncontrolled diabetes mellitus
12. Serious illness
13. Poor general health as judged by physician
14. Participation in concurrent clinical trials or previous trials within 3 months of screening
15. Previous treatment with ACT in the affected knee
16. Microfracture performed less than 1 year before screening in the affected knee
17. Alcohol or drug (medication) abuse
18. Meniscal transplant in the affected knee
19. Meniscal suture (in the affected knee) three months prior to baseline
20. Mosaicplasty (Osteoarticular Transplant System, OATS) in the affected knee
21. Having received hyaluronic acid intra-articular injections in the affected knee within the last 3 months before baseline
22. Taking specific osteoarthritis drugs such as chondroïtin sulfate, diacerein, nglucosamine,piascledine, capsaicin within 2 weeks before baseline
23. Corticosteroid treatment by systemic or intraarticular route within the last month of baseline or intramuscular or oral corticosteroïds within the last 2 weeks before baseline
24. Chronic use of anticoagulants
25. Any concomitant painful or disabling disease of the spine, hips or lower limbs that would interfere with evaluation of the afflicted knee
26. Any clinically significant or symptomatic vascular or neurological disorder of the lower extremities
27. Any evidence of the following diseases in the affected knee: septic arthritis, inflammatory joint disease, recurrent episodes of pseudogout, Paget's disease of bone, ochronosis, acromegaly, haemochromatosis, Wilson's disease, primary osteochondromatosis, heritable disorders, collagen gene mutation
28. Current diagnosis of osteomyelitis, human immunodeficiency virus (HIV-1,-2) and/or hepatitis C virus (HCV) infection

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 102 (Actual)
Dates: Start 2010-10; Primary Completion 2017-09 (Actual); Study Completion 2020-02 (Actual)

PRIMARY OUTCOMES:
Change of overall KOOS | 24 months after the end of the respective treatment
  Change of overall KOOS (Knee Injury and Osteoarthritis Outcome Score)from baseline (Day 0)to final assessment compared between ACT3D-CS (co.don chondrosphere) and MF (microfracture)

SECONDARY OUTCOMES:
Change of overall KOOS | 12, 36, 48, 60 months after the end of the respective treatment
  Change of overall KOOS(Knee Injury and Osteoarthritis Outcome Score) from baseline (Day 0) to 12 months, 36, 48, 60 months after the end of the respective treatment,compared between ACT3D-CS and MF
Change of the 5 subscores of the KOOS | 12, 24, 36, 48, 60 months after the end of the respective treatment
  Change of the 5 subscores of the KOOS (Pain, other Symptoms, Function in daily living (ADL), Function in sport and recreation (Sport/Rec), knee related Quality of life (QoL)) for both treatment groups compared between ACT3D-CS and MF
MOCART (MRI Score) | 12, 24, 36, 48 and 60 months after transplantation or microfracture
  MOCART (MRI Score) 12, 24, 36, 48 and 60 months after transplantation or microfracture compared between ACT3D-CS and MF
Arthroscopy and biopsy | 24 months
  Arthroscopy and biopsy at 24 months after transplantation/ microfracture, assessment of cartilage repair after ACT3D and microfracture to be compared between ACT3D-CS and MF
ICRS Visual Histological Assessment Score | 24 months after respective treatment
  ICRS Visual Histological Assessment Score at final assessment (24 months) compared between ACT3D-CS and MF
Bern Score and additional histological assessment scores | 24 months after the respective treatment
  Bern Score and additional histological assessment scores at final assessment (24 months) compared between ACT3D-CS and MF
Change of ICRS/IKDC | 12, 24, 36, 48 and 60 months after the end of the respective treatment
  Change of ICRS/IKDC from baseline (Day 0) to 12, 24, 36, 48 and 60 months after the end of the respective treatment, compared between ACT3D-CS and MF
Change of modified Lysholm Score | 12, 24, 36, 48 and 60 months after the end of the respective treatment
  Change of modified Lysholm Score from baseline (Day 0) to 12, 24, 36, 48 and 60 months after the end of the respective treatment compared between ACT3D-CS and MF
Days of absence from work (employment) and/or days of inability to follow usual activities | annual
  Days of absence from work (employment) and/or days of inability to follow usual activities during the last year or since the last visit, respectively, and time point when patient was back to work and/or to follow usual activities
Safety Parameters | 3,12,24 months after respective treatment
  Frequence and type of adverse Events Vital signs Physical examination Concomitant pain medication Laboratory parameters

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Fickert, Ph.D., Principal Investigator — Universitätsmedizin Mannheim
Locations (12):
- Germany (9):
  - Universitätsklinikum der Albert-Ludwig-Universität Freiburg, Department Othopädie und Traumatologie, Freiburg im Breisgau, Baden-Würrtemberg
  - Waldkrankenhaus "Rudolf Elle" GmbH Klinik für Orthopädie und Unfallchirurgie, Eisenberg, Tühringen
  - Gelenk-und Wirbelsäulenzentrum Steglitz, Berlin
  - DRK-Kliniken Westend, Berlin
  - St. Vinzenz-Hospital, Dinslaken
  - Orthopädische Klinik der Medizinischen Hochschule Hannover, Hanover
  - Lubinus Clinicum Kiel, Kiel
  - DRK Krankenhaus Luckenwalde, Luckenwalde
  - Orthopädisch-Unfallchirurgisches Zentrum, Mannheim
- Poland (3):
  - Uniwersytecki Szpital Kliniczny w Białymstoku, Bialystok
  - Wojewódzki Szpital Chirurgii Urazowej, Piekary Śląskie
  - Centrum Medycyny Sportowej, Warsaw

REFERENCES:
- [Derived] Hoburg A, Niemeyer P, Laute V, Zinser W, Becher C, Kolombe T, Fay J, Pietsch S, Kuzma T, Widuchowski W, Fickert S. Matrix-Associated Autologous Chondrocyte Implantation with Spheroid Technology Is Superior to Arthroscopic Microfracture at 36 Months Regarding Activities of Daily Living and Sporting Activities after Treatment. Cartilage. 2021 Dec;13(1_suppl):437S-448S. doi: 10.1177/1947603519897290. Epub 2020 Jan 1. PMID 31893951
- [Derived] Niemeyer P, Laute V, Zinser W, Becher C, Kolombe T, Fay J, Pietsch S, Kuzma T, Widuchowski W, Fickert S. A Prospective, Randomized, Open-Label, Multicenter, Phase III Noninferiority Trial to Compare the Clinical Efficacy of Matrix-Associated Autologous Chondrocyte Implantation With Spheroid Technology Versus Arthroscopic Microfracture for Cartilage Defects of the Knee. Orthop J Sports Med. 2019 Jul 10;7(7):2325967119854442. doi: 10.1177/2325967119854442. eCollection 2019 Jul. PMID 31317047